CLINICAL TRIAL: NCT00057590
Title: Outreach and Treatment for Depression in the Labor Force
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: R01MH061941 (NIH); R01MH061941 (NIH); DSIR 82-SEDX
Record Dates: First submitted 2003-04-04; First posted 2003-04-07 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

INTERVENTIONS:
Behavioral: Care manager outreach and monitoring

SUMMARY:
This study will assess the effects of depression treatment on employee productivity. This study will also evaluate the impact of depression screening and outreach on employees' receptivity to treatment.

DETAILED DESCRIPTION:
This study is conducted in three phases. In the first phase, employees from various companies participate in an on-line Health Risk Assessment survey at a secure website. Those who display symptoms of depression participate in a brief telephone interview to confirm the depression diagnosis.

In the second phase, depressed participants are randomly assigned to receive either intervention treatment or usual care for 18 months. The intervention consists of periodic telephone contact with a mental health clinician who provides education regarding depression and its treatment. Participants receiving the intervention are also provided with resources to obtain psychotherapy and/or pharmacotherapy. Those who do not seek treatment are monitored and supported. Participants in the usual care arm are informed of their possible depression and are encouraged to seek professional treatment.

The final phase of the study involves data analysis and dissemination of aggregated results. Surveys and questionnaires are used to assess participants.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive episode
* Employed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590
Dates: Start 2003-03

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard Medical School, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Wang PS, Simon GE, Avorn J, Azocar F, Ludman EJ, McCulloch J, Petukhova MZ, Kessler RC. Telephone screening, outreach, and care management for depressed workers and impact on clinical and work productivity outcomes: a randomized controlled trial. JAMA. 2007 Sep 26;298(12):1401-11. doi: 10.1001/jama.298.12.1401. PMID 17895456